CLINICAL TRIAL: NCT02348606
Title: A Twelve-Week, Double-Blind, Placebo-Controlled, Randomized, Parallel-Group, Multicenter Study of the Safety and Efficacy of JZP-110 [(R)-2-amino-3-phenylpropylcarbamate Hydrochloride] in the Treatment of Excessive Sleepiness in Subjects With Obstructive Sleep Apnea (OSA)
Brief Title: "Twelve-week Study of the Safety and Efficacy of JZP-110 in the Treatment of Excessive Sleepiness in OSA"
Acronym: OSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-003
Record Dates: First submitted 2015-01-15; First posted 2015-01-28 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 37.5 mg of JZP-110 (Active Comparator): Once Daily Dosing
  Interventions: Drug: JZP-110
- 75 mg of JZP-110 (Active Comparator): Once Daily Dosing
  Interventions: Drug: JZP-110
- 150 mg of JZP-110 (Active Comparator): Once Daily Dosing
  Interventions: Drug: JZP-110
- 300 mg of JZP-110 (Active Comparator): Once Daily Dosing
  Interventions: Drug: JZP-110
- Placebo (Active Comparator): Once Daily Dosing
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: JZP-110
  Arms: 150 mg of JZP-110; 300 mg of JZP-110; 37.5 mg of JZP-110; 75 mg of JZP-110
Drug: Placebo oral tablet
  Arms: Placebo

SUMMARY:
This trial is a 12 week, randomized, double-blind, placebo controlled, multicenter, 5-arm parallel group study of safety and efficacy of JZP-110 in the treatment of excessive sleepiness in adult subjects with OSA.

ELIGIBILITY:
Major Inclusion Criteria:

1. Male or female between 18 and 75 years of age, inclusive
2. Diagnosis of OSA according to ICSD-3 criteria
3. Body mass index from 18 to <45 kg/m2
4. Consent to use a medically acceptable method of contraception
5. Willing and able to provide written informed consent

Major Exclusion Criteria:

1. Female subjects who are pregnant, nursing, or lactating
2. Any other clinically relevant medical, behavioral, or psychiatric disorder other than OSA that is associated with excessive sleepiness
3. History or presence of bipolar disorder, bipolar related disorders, schizophrenia, schizophrenia spectrum disorders, or other psychotic disorders according to DSM-5 criteria
4. History or presence of any acutely unstable medical condition, behavioral or psychiatric disorder (including active suicidal ideation), or surgical history that could affect the safety of the subject or interfere with study efficacy, safety, PK assessments, or the ability of the subject to complete the trial per the judgment of the Investigator.
5. History of bariatric surgery within the past year or a history of any gastric bypass procedure
6. Presence or history of significant cardiovascular disease
7. Use of any over-the-counter (OTC) or prescription medications that could affect the evaluation of excessive sleepiness
8. Received an investigational drug in the past 30 days or five half-lives
9. Previous exposure to or participation in a clinical trial of JZP-110 (ADX-N05, R228060, or YKP10A)
10. History of phenylketonuria (PKU) or history of hypersensitivity to phenylalanine-derived products

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (59):
- United States (45):
  - Pulmonary Associates, Glendale, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - UC San Diego Medical Center, La Jolla, California
  - So Cal Institute For Respiratory Diseases, Inc., Los Angeles, California
  - Pacific Sleep Medicine, Oceanside, California
  - Stanford University Center for Narcolepsy, Redwood City, California
  - Pacific Research Network, Inc., San Diego, California
  - PAB Clinical Research, Brandon, Florida
  - MD Clinical, Hallandale, Florida
  - Clinical Research Group of St. Petersburg, St. Petersburg, Florida
  - Florida Pediatric Research Institute, Winter Park, Florida
  - NeuroTrials Research Inc., Atlanta, Georgia
  - SleepMed of Central Georgia, Macon, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Illinois at Chicago College of Nursing, Chicago, Illinois
  - Kentucky Research Group, Louisville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - The Center for Sleep & Wake Disorders, Chevy Chase, Maryland
  - Neurocare, Inc., Newton, Massachusetts
  - Henry Ford Hospital Sleep Disorders & Research Center, Detroit, Michigan
  - Clinical Neurophysiology Services, Sterling Heights, Michigan
  - Minnesota Lung Center, Edina, Minnesota
  - Sleep Medicine & Research Center, St. Luke's Hospital, Chesterfield, Missouri
  - University of Missouri, Columbia, Missouri
  - Clayton Sleep Institute, St Louis, Missouri
  - Clinilabs, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Hickory Research Center, Hickory, North Carolina
  - Hickory Research Center, ARSM Research, LLC, Huntersville, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Northcoast Clinical Trials Inc., Beachwood, Ohio
  - Sleep Management Institute, Cincinnati, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Southwest Cleveland Sleep Research Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Sleep Medicine & Neuroscience Institute, Dublin, Ohio
  - Mercy St. Anne & Mercy St. Charles Sleep Disorders Center, Toledo, Ohio
  - Sleep Med of South Carolina, Columbia, South Carolina
  - FutureSearch Trials of Neurology LP, Austin, Texas
  - Todd J. Swick, Houston, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas
  - Swedish Medical Center, Seattle, Washington
- Canada (5):
  - London Health Sciences Centre, London, Ontario
  - Niagra Clinical Research, Niagra Falls, Ontario
  - Toronto Sleep Institute, Toronto, Ontario
  - Toronto Psychiatric Research Foundation, Toronto, Ontario
  - Pediatric Sleep Research Inc., Toronto, Ontario
- France (3):
  - Hospital Roger Salengro, Lille
  - Universite Paris 5 Hôtel-Dieu, Paris
  - Hopital Bichat - Claude Bernard, Paris
- Germany (5):
  - medbo Bezirksklinikum Regensburg Schlafmedizinisches Zentrum, Regensburg, Bavaria
  - Universitätsklinikum Münster Department für Neurologie, Münster, North Rhine-Westphalia
  - Advanced Sleep Research GmbH, Berlin
  - Studienzentrum Wilhelmshoehe, Kassel
  - Somni bene GmbH Institut für Medizinische Forschung und Schlafmedizin Schwerin GmbH, Schwerin
- Sleep Wake Center SEIN Heemstede, Heemsteded, North Holland, Netherlands

REFERENCES:
- [Derived] Rosenberg R, Thorpy MJ, Dauvilliers Y, Schweitzer PK, Zammit G, Gotfried M, Bujanover S, Scheckner B, Malhotra A. Incidence and duration of common early-onset adverse events in randomized controlled trials of solriamfetol for treatment of excessive daytime sleepiness in obstructive sleep apnea and narcolepsy. J Clin Sleep Med. 2022 Jan 1;18(1):235-244. doi: 10.5664/jcsm.9550. PMID 34283019
- [Derived] Schweitzer PK, Mayer G, Rosenberg R, Malhotra A, Zammit GK, Gotfried M, Chandler P, Baladi M, Strohl KP. Randomized Controlled Trial of Solriamfetol for Excessive Daytime Sleepiness in OSA: An Analysis of Subgroups Adherent or Nonadherent to OSA Treatment. Chest. 2021 Jul;160(1):307-318. doi: 10.1016/j.chest.2021.02.033. Epub 2021 Feb 22. PMID 33631141
- [Derived] Weaver TE, Menno DM, Bron M, Crosby RD, Morris S, Mathias SD. Determination of thresholds for minimally important difference and clinically important response on the functional outcomes of sleep questionnaire short version in adults with narcolepsy or obstructive sleep apnea. Sleep Breath. 2021 Sep;25(3):1707-1715. doi: 10.1007/s11325-020-02270-3. Epub 2021 Jan 4. PMID 33394323
- [Derived] Rosenberg R, Baladi M, Bron M. Clinically relevant effects of solriamfetol on excessive daytime sleepiness: a posthoc analysis of the magnitude of change in clinical trials in adults with narcolepsy or obstructive sleep apnea. J Clin Sleep Med. 2021 Apr 1;17(4):711-717. doi: 10.5664/jcsm.9006. PMID 33226332
- [Derived] Weaver TE, Drake CL, Benes H, Stern T, Maynard J, Thein SG, Andry JM Sr, Hudson JD, Chen D, Carter LP, Bron M, Lee L, Black J, Bogan RK. Effects of Solriamfetol on Quality-of-Life Measures from a 12-Week Phase 3 Randomized Controlled Trial. Ann Am Thorac Soc. 2020 Aug;17(8):998-1007. doi: 10.1513/AnnalsATS.202002-136OC. PMID 32353246
- [Derived] Schweitzer PK, Rosenberg R, Zammit GK, Gotfried M, Chen D, Carter LP, Wang H, Lu Y, Black J, Malhotra A, Strohl KP; TONES 3 Study Investigators. Solriamfetol for Excessive Sleepiness in Obstructive Sleep Apnea (TONES 3). A Randomized Controlled Trial. Am J Respir Crit Care Med. 2019 Jun 1;199(11):1421-1431. doi: 10.1164/rccm.201806-1100OC. PMID 30521757

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Note: 476 subjects were enrolled and randomized, however 2 subjects never received drug. This resulted in 474 subjects comprising the safety population.
Pre-assignment Details: During screening, subjects completed a medical exam. An overnight Polysomnography (PSG) assessment followed by MWT and 24-hour ABPM were conducted at baseline. After successful completion of the screening and baseline visits subjects were randomized in a 1:1:2:2:2 ratio to receive 37.5, 75, 150, or 300 mg JZP- 110 or placebo.
Groups:
- 37.5 mg of JZP-110: 37.5 mg JZP-110 administered orally, once daily (QD), for the 12-week treatment phase.
- 75 mg of JZP-110: 75 mg JZP-110 administered orally, QD, for the 12-week treatment phase.
- 150 mg of JZP-110: Subjects randomized to receive 150 mg JZP-110 initially received 75 mg JZP-110 from Day 1 through Day 3 of the treatment phase, and received 150 mg JZP-110 starting on Day 4, administered orally, QD.
- 300 mg of JZP-110: Subjects randomized to receive 300 mg JZP-110 initially received 150 mg JZP-110 from Day 1 through Day 3 of the treatment phase and received 300 mg JZP-110 starting on Day 4, administered orally, QD.
- Placebo: Placebo administered orally, QD, for the 12 week treatment phase.
Period: Overall Study
Arm/Group | 37.5 mg of JZP-110 | 75 mg of JZP-110 | 150 mg of JZP-110 | 300 mg of JZP-110 | Placebo
Started | 58 | 62 | 117 | 118 | 119
Completed | 49 | 54 | 106 | 94 | 101
Not Completed | 9 | 8 | 11 | 24 | 18

BASELINE CHARACTERISTICS:
Groups:
- 37.5 mg of JZP-110: 37.5 mg JZP-110 administered orally, QD, for the 12-week treatment phase.
- Total: Total of all reporting groups
Arm/Group | 37.5 mg of JZP-110 | 75 mg of JZP-110 | 150 mg of JZP-110 | 300 mg of JZP-110 | Placebo | Total
Number analyzed (Participants) | 58 | 62 | 117 | 118 | 119 | 474
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (10.19) | 54.4 (11.46) | 52.7 (10.57) | 53.2 (10.62) | 54.1 (11.41) | 53.9 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 27 | 45 | 44 | 42 | 177
  Male | 39 | 35 | 72 | 74 | 77 | 297
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 3 | 1 | 3 | 6 | 4 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1 | 2
  Black or African American | 10 | 14 | 18 | 21 | 26 | 89
  White | 45 | 46 | 93 | 90 | 87 | 361
  More than one race | 0 | 1 | 2 | 1 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Maintenance of Wakefulness Test (MWT) From Baseline to Week 12
Description: Change in mean sleep latency time (in minutes) as determined from the first 4 trials of a 40-minute MWT from baseline to Week 12.
Time Frame: Baseline to Week 12
Population: Fifteen subjects in the Safety Population were excluded from the Modified Intent-to Treat (mITT) Population resulting in a total of 459 subjects.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | 37.5 mg of JZP-110 | 75 mg of JZP-110 | 150 mg of JZP-110 | 300 mg of JZP-110 | Placebo
Number analyzed (Participants) | 56 | 58 | 116 | 115 | 114
minutes | 4.74 (1.418) | 9.08 (1.358) | 10.96 (0.973) | 12.99 (1.038) | 0.21 (0.997)

2. Primary Outcome: Change in ESS Score From Baseline to Week 12
Description: Change in Epworth Sleepiness Scale (ESS) score from Baseline to Week 12. A negative change from baseline represents improvement in excessive sleepiness.
  The ESS is a self-administered questionnaire with 8 questions. Each activity is scored on a scale ranging from 0-3, with 0 = would never fall asleep, and 3 = high chance of falling asleep. The total score ranges from 0-24, with a higher number representing an increased propensity for sleepiness. An analysis of covariance (ANCOVA) was used for the analysis of ESS scores. The response variable was the change in ESS score from baseline.
Time Frame: Baseline to Week 12
Population: Fifteen subjects in the Safety Population were excluded from the mITT Population resulting in a total of 459 subjects.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | 37.5 mg of JZP-110 | 75 mg of JZP-110 | 150 mg of JZP-110 | 300 mg of JZP-110 | Placebo
Number analyzed (Participants) | 56 | 58 | 116 | 115 | 114
points on a scale | -5.1 (0.64) | -5.0 (0.62) | -7.7 (0.44) | -7.9 (0.46) | -3.3 (0.45)

3. Secondary Outcome: Subjects Reported Improved on the Patient Global Impression of Change (PGIc) at Week 12
Description: Percentage of subjects reported as improved (minimally, much, or very much) on the PGIc at Week 12. PGIc was rated by subjects and measures the change in their condition since start of treatment on a 7-point scale ranging from 1 = very much improved to 7 = very much worse.
  This is the key secondary endpoint.
Time Frame: 12 Weeks
Population: Fifteen subjects in the Safety Population were excluded from the mITT Population resulting in a total of 459 subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | 37.5 mg of JZP-110 | 75 mg of JZP-110 | 150 mg of JZP-110 | 300 mg of JZP-110 | Placebo
Number analyzed (Participants) | 56 | 58 | 116 | 115 | 114
percentage of subjects | 55.4 | 72.4 | 89.7 | 88.7 | 49.1

4. Secondary Outcome: Change in Sleep Latency Time on Each of the 5 MWT Trials at Week 12
Description: Time course of efficacy in MWT: Change in sleep latency (in minutes) on each of the 5 MWT trials at week 12.
Time Frame: Baseline and Week 12
Population: Fifteen subjects in the Safety Population were excluded from the mITT Population resulting in a total of 459 subjects.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | 37.5 mg of JZP-110 | 75 mg of JZP-110 | 150 mg of JZP-110 | 300 mg of JZP-110 | Placebo
Number analyzed (Participants) | 56 | 58 | 116 | 115 | 114
minutes
  Trial 1 | 3.03 (1.881) | 5.77 (1.808) | 10.87 (1.284) | 12.48 (1.401) | -0.40 (1.327)
  Trial 2 | 6.93 (1.928) | 9.47 (1.849) | 11.91 (1.332) | 14.94 (1.425) | -0.44 (1.380)
  Trial 3 | 3.59 (1.837) | 11.32 (1.751) | 11.50 (1.261) | 10.90 (1.340) | 0.58 (1.294)
  Trial 4 | 6.11 (1.845) | 9.04 (1.794) | 8.93 (1.272) | 11.94 (1.359) | 1.29 (1.305)
  Trial 5 | 3.57 (1.952) | 7.75 (1.839) | 8.05 (1.347) | 7.59 (1.432) | 0.18 (1.361)

5. Secondary Outcome: Change in the Mean Sleep Latency Time as Determined From the First 4 Trials of a 40-minute MWT From Baseline to Week 4
Description: Change in mean sleep latency time (in minutes) as determined from the first 4 trials of a 40-minute MWT from baseline to week 4.
Time Frame: Baseline to Week 4
Population: Fifteen subjects in the Safety Population were excluded from the mITT Population resulting in a total of 459 subjects.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | 37.5 mg of JZP-110 | 75 mg of JZP-110 | 150 mg of JZP-110 | 300 mg of JZP-110 | Placebo
Number analyzed (Participants) | 56 | 58 | 116 | 115 | 114
minutes | 4.53 (1.360) | 7.20 (1.307) | 11.69 (0.932) | 13.77 (0.976) | 1.24 (0.942)

6. Secondary Outcome: Change in ESS Score From Baseline to Week 1, Week 4, and Week 8
Description: Change in Epworth Sleepiness Scale (ESS) score from Baseline to Weeks 1, 4, and 8. A negative change from baseline represents improvement in excessive sleepiness.
  The ESS is a self-administered questionnaire with 8 questions. Each activity is scored on a scale ranging from 0-3, with 0 = would never fall asleep, and 3 = high chance of falling asleep. The total score ranges from 0-24, with a higher number representing an increased propensity for sleepiness. An analysis of covariance (ANCOVA) was used for the analysis of ESS scores. The response variable was the change in ESS score from baseline.
Time Frame: Baseline to Weeks 1, 4, and 8
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | 37.5 mg of JZP-110 | 75 mg of JZP-110 | 150 mg of JZP-110 | 300 mg of JZP-110 | Placebo
Number analyzed (Participants) | 56 | 58 | 116 | 115 | 114
points on a scale
  Week 1 | -4.5 (0.66) | -4.4 (0.65) | -5.5 (0.46) | -6.6 (0.46) | -2.6 (0.47)
  Week 4 | -4.7 (0.65) | -4.8 (0.63) | -6.1 (0.45) | -6.6 (0.46) | -2.9 (0.45)
  Week 8 | -4.7 (0.70) | -6.3 (0.67) | -6.9 (0.48) | -7.7 (0.50) | -3.8 (0.49)

7. Secondary Outcome: Percentage of Subjects Reported as Improved on the PGIc at Week 1, Week 4, and Week 8
Description: Percentage of subjects reported as improved (minimally, much, or very much) on the PGIc at Week 1, Week 4, and Week 8. PGIc was rated by subjects and measures the change in their condition since treatment start on a 7-point scale ranging from 1 = very much improved to 7 = very much worse.
Time Frame: Weeks 1, 4, and 8
Population: Fifteen subjects in the Safety Population were excluded from the mITT Population resulting in a total of 459 subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | 37.5 mg of JZP-110 | 75 mg of JZP-110 | 150 mg of JZP-110 | 300 mg of JZP-110 | Placebo
Number analyzed (Participants) | 56 | 58 | 116 | 115 | 114
percentage of subjects
  Week 1 | 58.9 | 65.5 | 78.3 | 82.5 | 47.4
  Week 4 | 60.7 | 77.6 | 84.5 | 84.3 | 53.5
  Week 8 | 57.1 | 79.3 | 88.8 | 87.8 | 57.0

8. Secondary Outcome: Percentage of Subjects Reported as Improved on the Clinical Global Impression of Change (CGIc) at Week 12
Description: Percentage of subjects reported as improved (minimally, much, or very much) on the CGIc at Week 12. CGIc was rated by clinicians and measures the change in the subject's condition since treatment starts on a 7-point scale ranging from 1= very much improved to 7= very much worse.
Time Frame: Week 12
Population: Fifteen subjects in the Safety Population were excluded from the mITT Population resulting in a total of 459 subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | 37.5 mg of JZP-110 | 75 mg of JZP-110 | 150 mg of JZP-110 | 300 mg of JZP-110 | Placebo
Number analyzed (Participants) | 56 | 58 | 116 | 115 | 114
percentage of subjects | 58.9 | 70.7 | 90.5 | 88.7 | 49.1

9. Secondary Outcome: Percentage of Subjects Reported as Improved on the CGIc at Week 1, Week 4, and Week 8
Description: Percentage of subjects reported as improved (minimally, much, or very much) on the CGIc at Week 1, Week 4, and Week 8. CGIc was rated by clinicians and measures the change in the subject's condition since treatment starts on a 7-point scale ranging from 1= very much improved to 7= very much worse.
Time Frame: Weeks 1, 4, and 8
Population: Fifteen subjects in the Safety Population were excluded from the mITT Population resulting in a total of 459 subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | 37.5 mg of JZP-110 | 75 mg of JZP-110 | 150 mg of JZP-110 | 300 mg of JZP-110 | Placebo
Number analyzed (Participants) | 56 | 58 | 116 | 115 | 114
percentage of subjects
  Week 1 | 62.5 | 60.3 | 75.7 | 82.6 | 46.5
  Week 4 | 60.7 | 77.6 | 85.2 | 81.7 | 52.6
  Week 8 | 55.4 | 74.1 | 87.8 | 87.8 | 49.1

ADVERSE EVENTS:
Time Frame: Through Week 14
Arm/Group | 37.5 mg of JZP-110 | 75 mg of JZP-110 | 150 mg of JZP-110 | 300 mg of JZP-110 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/62 | 0/117 | 0/118 | 0/119
Serious Adverse Events (participants affected / at risk) | 2/58 | 0/62 | 1/117 | 0/118 | 2/110
Other Adverse Events (participants affected / at risk) | 17/58 | 21/62 | 41/117 | 60/118 | 30/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 37.5 mg of JZP-110 (N=58) | 75 mg of JZP-110 (N=62) | 150 mg of JZP-110 (N=117) | 300 mg of JZP-110 (N=118) | Placebo (N=110)
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Streptococcal endocarditis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 37.5 mg of JZP-110 (N=58) | 75 mg of JZP-110 (N=62) | 150 mg of JZP-110 (N=117) | 300 mg of JZP-110 (N=118) | Placebo (N=119)
Headache (Nervous system disorders) | 4 | 5 | 10 | 17 | 10
Feeling jittery (General disorders) | 3 | 3 | 1 | 7 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 6 | 16 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 3 | 11 | 2
Irritability (Psychiatric disorders) | 3 | 0 | 4 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 10 | 12 | 7
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 5 | 8 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 5 | 9 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 9 | 14 | 1
Nasopharyngitis (Metabolism and nutrition disorders) | 2 | 1 | 7 | 8 | 8
Sinusitis (Metabolism and nutrition disorders) | 1 | 4 | 0 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review trial results communications prior to public release and can embargo such communications for a period of at least 60 days from the time submitted to sponsor for review. If requested by sponsor, the PI will withhold publication for up to an additional 30 days. Furthermore, the first publication of study results must be a joint publication of all study sites unless a joint manuscript has not been submitted for publication within 12 months of completion of the study.

DOCUMENTS (2):
  • Study Protocol (2016-02-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT02348606/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT02348606/SAP_001.pdf